CLINICAL TRIAL: NCT00782223
Title: Assessment of Hip, Spine and Lower Limbs Digital Radiograph Measurements in Pediatric Population: Using PACS Integrated Computer Software (TraumaCad From OrthoCrat)
Brief Title: Assessment of Digital Radiograph Measurements of Hip,Spine and Lower Limbs
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Tel-Aviv Sourasky Medical Center, Tel-Aviv Sourasky Medical Center
Other Study IDs: 0135-08-TLV
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: hips, spine, lower limb, digital radiograph measurements, TraumaCad, digital software; Measurements of orthopaedic parameters on digital X-rays using particular software

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1: Hip X-rays DDH
- 2: Hip X-rays, CP
- 3: Long standing lower Limb X-rays
- 4: Scoliosis, AP X-rays
- 5: Scoliosis Lateral X-rays

SUMMARY:
Research Protocol Assessment of Hip, Spine and Lower Limbs Digital Radiograph Measurements in Pediatric Population: using PACS integrated Computer Software (TraumaCad from OrthoCrat ™).

Introduction The integration of the PACS system into many medical institutions created a plethora of digital measurements to assess anatomic and deformity parameters for torso and limbs.

A number of commercial digital software is being offered to supply the medical practioner with tools to assess normal and pathological bony architecture land marks.

The relevant architecture of the pelvis (hip joint), spine and the length and alignment of lower limbs may be measured using these digital software's.

The validity and accuracy of digital work in comparison to conventional radiographs has been studied recently, mainly with lower extremity axial alignment, the digital length and anatomical angles measurements were found to be more reliable in terms of intra observer reliability than conventional radiographs (1, 2).

Study purposes

1. To compare the, accuracy and reliability of specifically designed digital software (TraumaCad from OrthoCrat ™) measurements using wizard guidance, to those produced by using the tool bar (ruler and angle guide tools) of the DICOM folder.
2. To assess intra and inter observer reliability of the TraumaCad software for different pediatric orthopaedics conditions.

   Methods *Twenty hip joins radiographs (AP views) of patients who suffer from Cerebral Palsy (10) and Developmental Dysplasia of the Hip (10) will be measured using the TraumaCad software hip joint wizard, and than again using basic tools of the DICOM folder.

   **Twenty spinal scoliosis radiographs (AP and Lat views) will be measured using the TraumaCad software templates.

   ***Ten digital radiographs of long leg standing (AP views) from normal and from patients with deformities will ne analyzed for length and angular differences using the LLD wizard.

   The following parameters will be measured *Hip joint radiographs: Acetabular Angle, Central Edge Angle, and Reimer's Index **Spinal radiographs: Cobe Angle (AP views), Coronal Balance, Sagital Balance. ***Long standing views: length of Femur and Tibia, mLDFA, mMPTA, mLDTA, JLCA, (the "Baltimore numbers").

   All measurements will be taken by 4 senior orthopaedic surgeons after consensus conference for the technique.

   Intra observer reliability will be tested by repeating the same set of measurements on 2 different dates, after all radiographs are randomly mixed and done at least 2 days apart. High resolution single computer will be used for all measurements by all participating surgeons.

   The intra and inter observer reliability for the hip joint measurements will be calculate to compared between TraumaCad software wizard and the DICOM measurements tools.

   All measurements using TraumaCad software will be analyzed for intra and inter observer reliability using accepted statistical tools.

   The study will be supervised by the department of statistics of TAU for maximum statistical significance.

1) Sailer J, Scharitzer M, Peloschek P, Giurea A, Imhof H, Grampp S.

Quantification of axial alignment of the lower extremity on conventional and digital total leg radiographs.

Eur Radiol. 2005 Jan; 15(1):170-3. Epub 2004 Aug 5.

2) Hankemeier S, Gosling T, Richter M, Hufner T, Hochhausen C, Krettek C.

Computer-assisted analysis of lower limb geometry: higher intraobserver reliability compared to conventional method.

Comput Aided Surg. 2006 Mar; 11(2):81-6

ELIGIBILITY:
Inclusion Criteria:

* hip, long leg & spine digital X-rays

Exclusion Criteria:

* inadequate X-rays

Ages: 2 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Digital X-rays from PACS system
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-12 (Estimated)